CLINICAL TRIAL: NCT00108849
Title: A 12 Month Double-blind, Randomized, Parallel-group, Placebo-controlled, Multi-center Trial to Investigate the Efficacy and Safety of Vagifem Low Dose (10 mcg 17beta-estradiol Vaginal Tablet) for the Treatment of Postmenopausal Atrophic Vaginitis Symptoms
Brief Title: Vagifem Low Dose for Postmenopausal Atrophic Vaginitis Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAG-2195
Record Dates: First submitted 2005-04-19; First posted 2005-04-20 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estradiol, 10 mcg

SUMMARY:
This trial is conducted in North America. The purpose of this study is to determine if Vagifem Low Dose is an effective and safe treatment for patients suffering from postmenopausal atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women whose last menstruation was at least two years previously

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2005-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms | after 12 months

SECONDARY OUTCOMES:
Objective parameters (vaginal Maturation Index/Value and vaginal pH)
Hyperplasia rate

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (53):
- United States (48):
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Carmichael, California
  - Novo Nordisk Investigational Site, Palo Alto, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Lakewood, Colorado
  - Novo Nordisk Investigational Site, New London, Connecticut
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Daytona Beach, Florida
  - Novo Nordisk Investigational Site, Palm Springs, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Alpharetta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Laurel, Maryland
  - Novo Nordisk Investigational Site, Lincoln, Nebraska
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Moorestown, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Mount Airy, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Eugene, Oregon
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, West Reading, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Jackson, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Sandy City, Utah
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (5):
  - Novo Nordisk Investigational Site, Kingston
  - Novo Nordisk Investigational Site, Montreal
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Toronto
  - Novo Nordisk Investigational Site, Winnipeg

REFERENCES:
- [Result] Mettler L, Olsen PG. Long-term treatment of atrophic vaginitis with low-dose oestradiol vaginal tablets. Maturitas. 1991 Dec;14(1):23-31. doi: 10.1016/0378-5122(91)90144-f. PMID 1791769
- [Derived] Derzko CM, Rohrich S, Panay N. Does age at the start of treatment for vaginal atrophy predict response to vaginal estrogen therapy? Post hoc analysis of data from a randomized clinical trial involving 205 women treated with 10 mug estradiol vaginal tablets. Menopause. 2020 Oct 5;28(2):113-118. doi: 10.1097/GME.0000000000001666. PMID 33038141
- [Derived] Simon J, Nachtigall L, Ulrich LG, Eugster-Hausmann M, Gut R. Endometrial safety of ultra-low-dose estradiol vaginal tablets. Obstet Gynecol. 2010 Oct;116(4):876-883. doi: 10.1097/AOG.0b013e3181f386bb. PMID 20859151
- [Derived] Simon J, Nachtigall L, Gut R, Lang E, Archer DF, Utian W. Effective treatment of vaginal atrophy with an ultra-low-dose estradiol vaginal tablet. Obstet Gynecol. 2008 Nov;112(5):1053-60. doi: 10.1097/AOG.0b013e31818aa7c3. PMID 18978105
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com